CLINICAL TRIAL: NCT01280851
Title: Comprehensive Morphological and Functional Assessment of Living Renal Donor With Magnetic Resonance Imaging With Comparison to Computed Tomographic Angiography and Renal Scintigraphy
Brief Title: Living Renal Donor MRI Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Kartik Jhaveri, University Health Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UHN10-0202-A
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Living Renal Donor
Keywords: Living renal donor; Magnetic Resonance Imaging; Renal vascular anatomy; Renal function
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — 1 hour of MRI exam will be performed in addition to the standard of care procedures, using low dose of gadolinium-based contrast (not investigational drug).

SUMMARY:
Accurate preoperative evaluation of a potential living renal donor's anatomy, vasculature and function is crucial to ensure optimal outcomes for both kidney donor and recipient in transplantation.

Currently abdominal ultrasound and spiral CT angiography are used to evaluate renal anatomy and vascular status, and renal scintigraphy to evaluate renal function. This imaging protocol exposes this relatively young and healthy population to a high radiation dose and potentially nephrotoxic contrast agents.

The investigators hypothesize that a single MR-based examination in the preoperative evaluation of potential kidney donor is a faster, safer, more cost effective and as accurate as the current multiple imaging work-up protocol.

DETAILED DESCRIPTION:
An accurate preoperative assessment of the renal donor is essential to minimize the risks for the donor & optimize the results for the recipient.

The current preoperative assessment includes Ultrasound, CT & Renal Scintigraphy. The latter two tests subjects the patient to the risk of a high radiation dose. Moreover, the use of iodinated contrast media during CT angiography may increase the risk of renal & systemic toxicity.

MRI can be a "one-stop shop" modality for preoperative assessment of living kidney donors. MRI also eliminates radiation exposure and the injection of potentially nephrotoxic iodinated contrast material.

The purpose of this study is to test the feasibility and evaluate the accuracy of a single MR-based examination, allowing for the comprehensive assessment of renal anatomy, function and vascular status in potential live kidney donors.

ELIGIBILITY:
Inclusion Criteria:

* Potential renal donors with no known renal disease (initial medical screening performed and scheduled for further imaging evaluation as renal donor);
* Age 18-65 years;
* No medications (birth control pills and vitamins are acceptable).

Exclusion Criteria:

* Pregnancy;
* Age <18 years or >65 years;
* MRI contrast allergy, general contraindications to MRI such as pacemaker, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Accuracy of MRI exam in kidney donors | 2 years
  To evaluate the accuracy of comprehensive Renal Magnetic Resonance Imaging (MRI) examination compared to CT angiography and Renal scintigraphy for the assessment of renal vascular anatomy and function in potential kidney donors.

SECONDARY OUTCOMES:
cost analysis | 2 years
  To perform a cost-analysis study to determine feasibility of replacing US, CT and Nuclear Scintigraphy by single MRI examination

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Jhaveri, MD, Principal Investigator — University Health Network, Toronto